CLINICAL TRIAL: NCT05006157
Title: Safety and Efficacy of the ViaOne Device for Pericardial Access - a Feasibility Study
Brief Title: Pericardial Access With ViaOne Device
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CardioVia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAV-CL-011
Record Dates: First submitted 2021-04-20; First posted 2021-08-16 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pericardial Access
Keywords: Pericardial space; pericardial access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ViaOne device (Experimental): ViaOne device will be used for percutaneous subxiphoid pericardial access utilizing a proprietary mechanism of entry into the pericardial sac
  Interventions: Device: ViaOne device

INTERVENTIONS:
Device: ViaOne device — ViaOne device is designed to allow percutaneous subxiphoid pericardial access utilizing a proprietary mechanism of entry into the pericardial sac.

SUMMARY:
ViaOne device is a tool designed to allow percutaneous subxiphoid pericardial access utilizing a proprietary mechanism of entry into the pericardial sac. In this study ViaOne will be used to obtain pericardial access in patients in whom electrophysiological diagnostic (mapping) and/or therapeutic (ablation) of epicardial sites via percutaneous subxiphoid approach to the to the normal, non-distended pericardial space is indicated.

DETAILED DESCRIPTION:
The primary objective of the study is to provide evidence of safety of ViaOne in obtaining percutaneous subxiphoid approach to the pericardial space. The secondary objective is to provide initial estimate of efficacy of ViaOne in obtaining percutaneous subxiphoid approach to the pericardial space.

Screening procedures will include laboratory analyses of the complete blood count, serum chemistry, coagulation parameters, and urine or serum ß-HCG test.A physical examination and collection of vital signs will be conducted. Medical history data and information on concomitant medications will be collected.

Once eligibility is verified, subjects will be scheduled for a procedure during which percutaneous subxiphoid pericardial access will be obtained using the ViaOne and its associated procedure. Time period between the study device insertion through the subxiphoid incision and guidewire insertion into the pericardial sac, overall time in procedure, and any procedural complications and device deficiencies will be recorded.

Follow-up visit will be conducted as part of the planned protocol procedures at up 5 ± 1 days after the procedure or at the time of discharge, whichever comes first. The visit will include evaluation of any adverse events and complications. Length of hospital stay will be recorded, where the discharge precedes or coincides with the final follow-up visit of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21
2. Electrophysiological diagnostic (mapping) and/or therapeutic (ablation) of epicardial sites via percutaneous subxiphoid approach to the to the normal, non-distended ericardial space is indicated.
3. Pre-treatment coagulation values within the following limits:

   * international normalized ratio 0.8 - 1.2
   * partial thromboplastin time 25 - 35''
4. Pre-treatment hematology and biochemistry values within the following limits:

   * hemoglobin ≥ 10 g/dL (g/100 mL)
   * platelets ≥ 150 x 10^9/L (x 10^3/mm^3)
   * white blood cells ≥ 3.0 x 10^9/L (x 10^3/mm^3)
   * absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1.5 x 10^3/mm^3)
   * serum creatinine < 1.5 mg/dL
   * aspartate aminotransferase < 1.5 x ULN (upper limit of norm)
   * alanine aminotransferase < 1.5 x ULN
   * alkaline phosphatase < 1.5 x ULN
5. Signed informed consent.

Exclusion Criteria:

* History of cardiac or pericardial surgery or prior pericardial ablation.
* History of chronic pericarditis.
* Known pericardial fibrosis and/or adhesions.
* Any anomaly in the chest anatomy.
* Myocardial infarction, past or present.
* Bleeding disorders.
* Hepatic enlargement.
* BMI > 40
* Participation in another interventional trial.
* Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of ViaOne device | through study completion, an average of 5 days
  Incidence of device-related adverse events through study completion, an average of 5 days

SECONDARY OUTCOMES:
Initial Efficacy of ViaOne device | through study completion, an average of 5 days
  Rate of success of pericardial space access, defined as guidewire insertion into the pericardial space.

CONTACTS AND LOCATIONS:
Overall Officials: David Luria, Principal Investigator — Hadassah MC, Jerusalem, Israel
Locations (4):
- Israel (2):
  - Hadassah Ein Kerem MC, Jerusalem
  - Shaare Zedek MC, Jerusalem
- Poland (2):
  - SzpitalKlinicznyPrzemienieniaPańskiegoUniwersytetuMedycznegoim. Karola Marcinkowskiego w Poznaniu, Poznan
  - MedicoverOpiekaSzpitalna, AlejaRzeczypospolitej 5, 02-972, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derejko P, Dzwonkowska D, Wrobel K, Kusnierz J, Bardyszewski A, Menshes Z, Hazan O, Leon A, Luria D, Lakkireddy D. Safety and Efficacy of a Novel Blunt-Tip Concealed-Needle Epicardial Access Device: First-in-Human Feasibility Study. JACC Clin Electrophysiol. 2022 Jul;8(7):908-912. doi: 10.1016/j.jacep.2022.04.016. Epub 2022 Apr 30. PMID 35750622